CLINICAL TRIAL: NCT07156773
Title: Study on Safety and Clinical Efficacy of XJN010 Nasal Spray in Patients With Parkinson's Disease Experiencing Off Episodes
Brief Title: The Study is Being Conducted to Evaluate the Safety and Efficacy of XJN010 Nasal Spray in Patients With Parkinson's Disease Experiencing Off Episodes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Novaken Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-Ⅱ-ZXDB-02
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XJN010 Nasal Spray (Experimental): The drug used is XJN010 Nasal Spray.
  Interventions: Drug: XJN010 Nasal Spray
- XJN010 Nasal Spray blank preparation. (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XJN010 Nasal Spray — In the XJN010 Nasal Spray group, subjects will receive XJN010 Nasal Spray，Based on the frequency of the "off" periods experienced by Parkinson's patients.
  Arms: XJN010 Nasal Spray
Drug: Placebo — In the XJN010 Nasal Spray blank preparation group, subjects will receive XJN010 Nasal Spray blank preparation, Based on the frequency of the "off" periods experienced by Parkinson's patients .
  Arms: XJN010 Nasal Spray blank preparation.

SUMMARY:
The study is being conducted to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of XJN010 Nasal Spray in Patients with Parkinson's Disease Experiencing Off Episodes

DETAILED DESCRIPTION:
A multi-center, randomized, double-blind, placebo-controlled trial design was adopted. Qualified subjects will be selected and enter the treatment period (D1 to D14). A total of 84 patients were included, and they were randomly assigned to the nasal spray group or the placebo group in a ratio of 3:1:3:1:3:1.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 30 to 85 years (inclusive);
* Diagnosed with Parkinson's disease according to the Chinese Diagnostic Criteria for Parkinson's Disease (2016), with a disease duration of at least 3 years;
* Patients with a Hoehn-Yahr stage rating (during "on" periods) of 1 to 3;
* Demonstrates responsiveness to levodopa (≥30% improvement/decrease in UPDRS-III score (motor examination) from "off" to "on" state following morning administration of routine levodopa dose);
* Patients must have no plans for conception from 2 weeks before the first dose until 1 month after the last dose, no plans to donate sperm, and agree to use highly effective contraception methods;
* Patients are capable of understanding the study requirements, voluntarily provide written informed consent, and are able to complete the study in compliance with the trial protocol.

Exclusion Criteria:

* Individuals with motor impairments that severely affect their ability to participate in and perform study procedures;
* Those exhibiting dyskinesia that significantly impacts daily functioning;
* Known hypersensitivity/allergic reaction or intolerance to any component of the investigational drug;
* Previous Parkinson's disease (PD) surgery (including but not limited to deep brain stimulation or brain cell transplantation) or planned PD surgery during the trial period;
* History of malignancy within the past 5 years, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, or ductal carcinoma in situ of the breast treated with radical surgery;
* History of severe psychiatric disorders within the past year, such as major depression, mania, schizophrenia, or patients with suicidal tendencies;
* Patients deemed unsuitable for intranasal administration by the investigator (e.g., severe rhinitis, nasal deformities, etc.);
* Those currently receiving centrally nervous system-active medications (e.g., sedatives, hypnotics, antidepressants, anxiolytics), except for those who have maintained a stable dose for at least 30 days prior to screening and can remain stable during the study;
* History of orthostatic hypotension or clinically significant hypotension or orthostatic hypotension identified during screening (orthostatic hypotension is defined as a drop in systolic blood pressure ≥20 mmHg or diastolic blood pressure ≥10 mmHg within 3 minutes of standing from a supine position)
* Any laboratory test during screening meeting the following criteria:

Liver function: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN); or total bilirubin >2 × ULN; Renal function: Serum creatinine >178 μmol/L;11. Pregnant or lactating females, or those with a positive pregnancy test during screening;

* History of drug or alcohol abuse within the past year;
* Participation in a clinical trial and use of an investigational drug within 1 month prior to screening or within 5 drug half-lives (whichever is longer);
* Any other condition considered by the investigator to make the patient unsuitable for participation in the trial.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS part III score | Day14
  MDS - Unified Parkinson's Disease Rating Scale Part III，The minimum score is 0 and the maximum is 4， higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The proportion of patients whose condition progresses from the "OFF" phase to the "on" phase and remains in the "on" phase state | Day14
  The proportion of patients whose condition progresses from the "closed" phase to the "open" phase and remains in the "open" phase state
The duration of the "OFF" period compared to the baseline value | Day14
  The duration of the "OFF" period compared to the baseline value
PDQ-39 score | Day14
  Parkinson's disease Questionnaire-39 score，The minimum score is 0 and the maximum is 4， higher scores mean a worse outcome.
Maximum blood concentration (Cmax) | 0 to 4 hour after administration
  Maximum blood concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University (Guangzhou Overseas Chinese Hospital), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a signed data sharing agreement.
Supporting Information: ICF
Time Frame: Data are available 6 months after the primary publication
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.novaken.cn/